CLINICAL TRIAL: NCT06571903
Title: Video-based Learning for Basic Surgical Skills - a Randomized Trial
Brief Title: Video-based Learning for Basic Surgical Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VBSS
Record Dates: First submitted 2024-07-11; First posted 2024-08-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Teaching Basic Surgical Techniques
Keywords: Video-based Learning; Basic Surgical Skills; mOSATS; Surgical Education; Teaching Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional Learning (No Intervention): Teaching with an expert tutor, in a in-person course
- Video-based Learning (Experimental): Teaching with videos for autonomous learning and practice
  Interventions: Other: Teaching from videos

INTERVENTIONS:
Other: Teaching from videos — Teaching from videos for independent study
  Arms: Video-based Learning

SUMMARY:
This is a prospective randomized study, intended to evaluate the effectiveness of teaching basic surgical techniques through video, comparing the results with those of traditional teaching

ELIGIBILITY:
Inclusion Criteria:

* Students from the 1st to 3rd years of the Integrated Master's Degree in Medicine at the University of Porto,
* Able to participate in a course of basic surgical techniques (simple suturing, X-stitches, U-stitches and Donatti points)

Exclusion Criteria:

* Participants is to have had prior contact with techniques surgical and/or minor surgery,
* Participants had contact with techniques surgical and/or minor surgery in the period between recruitment and completion of the proposed learning

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the qualities of the techniques (Objective Structured Assessment of Technical Skills (OSATS) modified scale) | 2 weeks
  Evaluate the quality of execution of the technical gesture and its retention on each group (teaching basic surgical techniques through video and traditional education (courses face-to-face)). The Objective Structured Assessment of Technical Skills (OSATS) modified scale is scored from 8 (worst performance) to 40 (best performance).
Time the participants took to complete the procedure | 2 weeks
  Time in minutes and seconds (mm:ss) that the participants took to complete the procedure on each group (teaching basic surgical techniques through video and traditional education (courses face-to-face)).

SECONDARY OUTCOMES:
Assessment of participants' involvement and interest (time of self-study in hours) | 1 month
  Time of self-study in hours and minutes (hh:mm), to check participants' involvement and interest in the teaching method through video.
Participant satisfaction with teaching method (Likert-like satisfaction questionnaire) | 1 day
  Likert-like satisfaction questionnaire scored from 5 (worst outcome) to 25 (best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Vitor Lopes, MD, PhD, Study Director — Faculty of Medicine of University of Porto
Locations (1):
- Faculty of Medicine of University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No